

# Effects of unilateral, bilateral and combined resistance training on the speed and accuracy of the serve in youth tennis players

| Expert Information | |
|---|---|
| Work Unit: | University of Putra Malaysia |
| Full name: | Ma Xudong |
| Title: | Effects of unilateral, bilateral and combined resistance |
| | training on the speed and accuracy of the serve in youth |
| | tennis players |
| Research Area: | Physical Education |
| Working Experience: | School assistant, coach |

#### Dear Professor,

My name is Ma Xudong, and I am a PhD student majoring in Physical education at Universiti Putra Malaysia (UPM). The aim of this study was to investigate the effects of single, bilateral and combined resistance training on the speed and accuracy of serving in Chinese amateur teenage tennis players. The subjects were young male tennis players aged 16-20 years from four universities in Gansu Province. The data obtained in this survey were used for academic research only. Therefore, I invited experts to evaluate and score the experimental design to help me better complete this experiment. Thank you very much.

The study was divided into control group (CG), experiment group 1 (EG1-unilateral group), experiment group 2 (EG2-bilateral group) and experiment group 3 (EG3-combined group). Used to compare the effects of different forms of resistance training on serve speed and accuracy. Previous studies have shown that unilateral and bilateral resistance training can effectively improve athletes' strength, explosive power, and speed (Speirs, et al., 2016; Davo, Jimenez, & Solana,., 2018), there is still controversy when comparing the advantages and disadvantages of two forms of resistance training (Ramirez-Campillo et al., 2015; Donathb & Wahl., 2022). In this study, unilateral resistance training, bilateral resistance training, and combined unilateral and bilateral resistance training were used as intervention modalities.

Based on the literature review, the training frequency of this experiment was arranged as 2 sessions/week, and the total training time was 6 weeks, with a fixed duration of each training session. Each training session lasted a maximum of 60 minutes. In this experiment, the interval between two

weekly training sessions was at least 24 h to prevent subjects from being in a fatigued state in the relevant muscle groups of the body and affecting the experimental level.

# 1. Pre-activation Prescription

| week | Intensity of Pre-activation | Type of<br>Warm-up | Type of Exercise | Intensity & Repetition | Sets | Recovery<br>Time |
|---|---|---|---|---|---|---|
| | CG | Routine<br>Warm-up | Routine Warm-up | NO | NO | NO |
| | EG1 | Dynamic<br>Warm-up | Dynamic warm<br>up<br>(Table1) | NO | | |
| 1-6 | EG2 | Dynamic<br>Warm-up | Dynamic<br>Warm-up<br>(Table1) | NO | 1 | 1min |
| | EG3 | Dynamic<br>Warm-up | Dynamic<br>Warm-up<br>(Table1) | NO | | |

#### Table1

| EG1 | EG2 | EG3 |
|------------------------|-----|-----|
| Dynamic Warm-Up (Time) | | |

- 1. High-knee walk. While walking, lift knee towards chest, raise body on toes, and swing alternating arms.
- 2. Straight-leg march. While walking with both arms extended in front of body, lift one extended leg towards hands then return to starting position before repeating with other leg.
- 3. Hand walk. With hands and feet on the ground and limbs extended, walk feet towards hands while keeping legs extended then walk hands forward while keeping limbs extended.
- 4. Lunge walks. Lunge forward with alternating legs while keeping torso vertical.
- 5. Backward lunge. Move backwards by reaching each leg as far back as possible.
- 6. High-knee skip. While skipping, emphasize height, highknee lift, and arm action.
- 7. Lateral shufflfle. Move laterally quickly without crossing feet.
- 8. Back pedal. While keeping feet under hips, take small steps to move backwards rapidly.
- 9. Heel-ups. Rapidly kick heels towards buttocks while moving forward.
- 10. High-knee run. Emphasize knee lift and arm swing while moving forward quickly.

This study recommends a warm-up with dynamic exercises and a cool-down using body stretching. Warm-up programmes have been shown to be effective in improving jumping performance and are recommended for young people as a standardised warm-up prior to RT (Faigenbaum et al., 2005).

Expert score: your evaluation of measurements is (the full score is 10 points, 9-10 points are very applicable, 7.5-8.5 points are applicable, 6-7 points are less applicable, and 4.5-5.5 points are not applicable.)

| Order | Items | Score |
|------------|---------------------------------------|-------|
| 1 | The Content of whole Training Program | |
| 2 | Intensity of Pre-activation | |
| 3 | Type of Warm-up | |
| 4 | Type of Exercise | |
| 5 | Intensity & Repetition | |
| 6 | Training Sets | |
| 6 | Recovery Time | |
| 3.5. 11.00 | 1 0 1 07 | 1 |

Modification Suggestions of Experts:

# 2. Basic Training Program

| EG1 | EG2 | EG3 | CG | |
|---|---|---|---|---|
| Dynamic W | /arm-Up and Training | | Routine Warm-Up and Training | |
| | | | | (Time) |
| High-knee walk- 1 | time (1min) | | • | Jogging - 1 time (10 min) |
| Straight-leg march | n -1 times (1min) | | • | traditional training (50min) |
| Hand walk - 1sets- | • Hand walk - 1sets- 1 time (1min) | | | Total time (60min) |
| • Lunge walks - 1 tir | me (1min) | | | |
| Backward lunge - | 1 time (1min) | | | |
| ● High-knee skip -1 | time (1min) | | | |
| Lateral shufflfle- 1 | time (1min) | | | |
| Back pedal -1 time | e (1min) | | | |
| Heel-ups -1 time ( | 1min ) | | | |
| ● High-knee run -1 t | time (1min) | | | |
| • Unilateral, bilateral, | combined resistance train | ning ( EG1, EG2, | | |
| EG3) (50 min) | | | | |
| • Total time (60min) | | | | |
| Training Content | Training Content | | | |
| (Training base phase (first two weeks): 65-75% of intensity, 2sets, 8raps) (NSCA, 2009) | | | | |

# Specific Intervention Prescription

## Unilateral resistance training programme

| Category | Free weight resistance training | Intervals | Rapid Contraction resistance |
|---|---|---|---|
| | movements | | Training |
| | (NSCA, 2009) | | (Carter, 2014) |
| Upper<br>limb | Unilateral Bench Press Dumbbell dominant limb: 50% 1RM, 4 × 8; Non-dominant limb: 50% 1RM, 4 × 8 VIPR energy barrel for unilateral bench press dominant limb: 50% 1RM, 4 × 8; Non-dominant limb: 50% 1RM, 4 × 8 | 2min | One-handed push-ups on box (dominant limb: 4 x 10; non-dominant limb: 4 x 10) medicine ball forward throw (dominant limb: 4 x 10; non-dominant limb: 4 x 10.) Stretch band continuous tennis swing action (dominant limb: 4 x 20; non-dominant limb: 4 x 20.) |
| lower limb | Bulgarian Arrow Squat dominant limb:50% 1RM, 4×8 Non-dominant limb:50% 1RM, 4×8 Bulgarian unilateral heel lift dominant limb:50% 1RM, 4 x 8 Non-dominant limb:50% 1RM, 4 x 8 | 2min | Self-weighted cross lunge jump (dominant limb: 4 x 10; non-dominant limb: 4 x 10) Single foot hurdle vertical jump 0.25cm (dominant limb: 4 x10; non-dominant limb: 4 x10) |
| | limb | Category movements (NSCA, 2009) Unilateral Bench Press Dumbbell dominant limb: 50% 1RM, 4 × 8; Non-dominant limb: 50% 1RM, 4 × 8 Upper limb VIPR energy barrel for unilateral bench press dominant limb: 50% 1RM, 4 × 8; Non-dominant limb: 50% 1RM, 4 × 8 Non-dominant limb: 50% 1RM, 4 × 8 lower limb Bulgarian unilateral heel lift dominant limb: 50% 1RM, 4 × 8 | Category movements (NSCA, 2009) Unilateral Bench Press Dumbbell dominant limb: 50% 1RM, 4 × 8; Non-dominant limb: 50% 1RM, 4 × 8 Upper limb VIPR energy barrel for unilateral bench press dominant limb: 50% 1RM, 4 × 8; Non-dominant limb: 50% 1RM, 4 × 8 Non-dominant limb: 50% 1RM, 4 × 8 Non-dominant limb: 50% 1RM, 4×8 Non-dominant limb: 50% 1RM, 4×8 Non-dominant limb: 50% 1RM, 4×8 Non-dominant limb: 50% 1RM, 4×8 2min Bulgarian unilateral heel lift dominant limb: 50% 1RM, 4 x 8 |

(Training base phase (first two weeks): 65-75% of intensity, 2sets, 8raps) (NSCA, 2009)

## Bilateral resistance training programme

| | Category | Free weight resistance training movements (NSCA, 2009) | Intervals | Rapid Contraction resistance Training (Carter, 2014) |
|---|---|---|---|---|
| Bilateral training (1h) | Upper<br>limb | Bench Press for Dumbbell (80-85%1RM 4×8) VIPR energy barrel for bench press (80-85%1RM 4×8) | 2min | High five with push-ups (4×10) Double-sided medicine ball forward throw (4×10) Stretch band continuous tennis swing action (Bilateral ) (4×20) |
| | lower limb | Bilateral Weight Squat (80-85%1RM 4×8) Bulgarian Heel Lift (80-85%1RM 4×8) | 2min | Jump box (3×10) Hurdle Vertical Jump 0.25cm, 4×10 |

(Training base phase (first two weeks): 65-75% of intensity, 2sets, 8raps) (NSCA, 2009)

## Combined (UL+BL) resistance training programme

| | Category | Free weight resistance training movements (NSCA, 2009) | Intervals | Rapid Contraction resistance Training (Carter, 2014) |
|---|---|---|---|---|
| Combined (UL+BL) Itraining (1h) | Upper<br>limb | Unilateral Bench Press Dumbbell dominant limb: 50% 1RM, 4 × 8; Non-dominant limb: 50% 1RM, 4 × 8 VIPR energy barrel for bench press (80-85%1RM 4×8) | 2min | One-handed push-ups on box (dominant limb: 4 x 10; non-dominant limb: 4 x 10) Double-sided medicine ball forward throw (4×10) Stretch band continuous tennis swing action (Bilateral and Unilateral) (2×20/2×20) |
| Co | lower limb | Bulgarian Arrow Squat dominant limb:50% 1RM, 4×8 Non-dominant limb:50% 1RM,4×8 Bulgarian Heel Lift (80-85%1RM 4×8) | 2min | Self-weighted cross lunge jump (dominant limb: 4x 10; non-dominant limb: 4 x 10) Hurdle Vertical Jump 0.25cm, 4×10 |

(Training base phase (first two weeks): 65-75% of intensity, 2sets, 8raps) (NSCA, 2009)

Expert score: your evaluation of training program is (the full score is 10 points, 9-10 points are very applicable, 7.5-8.5 points are applicable, 6-7 points are less applicable, and 4.5-5.5 points are not applicable.)

| Order | Items | Score |
|-------|---------------------------------------|-------|
| 1 | The Content of whole Training Program | |
| 2 | Warm-up | |
| 3 | Training Duration & Frequency | |
| 4 | Type of Exercise | |
| 5 | Training Intensity & Repetition | |
| 6 | Training Sets | |
| 7 | Recovery Time | |

## 3.Instruments

#### Sport performance tests (The contribution of the tennis serve)

| TEST | 5RM-BS | 5RM-BP | CMJ | OMB | SJF | SRT | HEC |
|---|---|---|---|---|---|---|---|
| PURPOSE | Maximum strength of the upper limb | Maximum strength of the lower limb | Maximum power of the lower limb | Maximum power of the upper limb | Flexibility of upper limb joints | Flexibility of lower limb joints | body coordination |
| EQUI<br>PAM | Barbell (kg) | Barbell (kg) | APP (cm) | Measuring tape (m) | Ruler with scale (cm) | Ruler with scale (cm) | Stop watch (times) |
| POSITION | Subjects were supine on a bench, which was parallel to the floor. The back of the subject should be close to the surface of the table, with the knees in the same direction as the toes | Subjects were instructed to<br>stand behind the barbell with<br>their feet shoulder-width apart<br>and their knees facing in the<br>same direction as their toes | The subject remains standing | The subject remains standing | Subjects remain standing | The subject remained in a seated position | The subject stood with a tennis ball in hand |
| ACTION | The subject held the dumbbell tightly. Subjects had to reach the specified depth with downward motion (90° at the elbow). In addition, the direction of the dumbbell should be consistent with the direction of the nipple throughout the movement | Move your toes outward 30°. The barbell was clenched and the hands rested on the scapula. The subject must reach the specified depth ((90° knee Angle)) when moving down. | The subjects kept their hands still and completed the jump during the squat | Subjects grabbed<br>the medicine ball<br>and threw it as<br>far as they could<br>over their heads | The upper limbs of<br>the subjects were<br>extended and<br>rotated backward<br>without tilting the<br>trunk | Subjects had<br>their legs<br>straight and<br>their upper<br>limbs<br>extended<br>forward | The subject threw the tennis ball against the wall and repeated the action until the ball fell to the ground |
| MEASUR<br>EMENT | The maximum weight that can be pushed | The maximum weight that can be pushed | The vertical height of the jump | Horizontal distance | The distance between the hands | Horizontal<br>distance | Number of times in 30 seconds |

#### Tennis serve performance

| Tennis serve performance | | |
|---|---|---|
| TEST | SPEED TEST | ACCURACY TEST |
| PURPOSE | Measure the speed of a tennis serve | To measure the accuracy of a tennis serve |
| EQUIPAMENT | radar gun (Bushnell-10-1911) | Figure 1 (score) |
| POSITION | The subject was prepared to complete the serve movement | The subject was prepared to complete the serve movement |
| ACTION | The subject completed the serve movement | The subject completed the serve movement |
| MEASUREMENT | Km/h | Score |



Figure 1-Tennis accuracy Tes

Expert score: your evaluation of measurements is (the full score is 10 points, 9-10 points are very applicable, 7.5-8.5 points are applicable, 6-7 points are less applicable, and 4.5-5.5 points are not applicable.)

| Order | Items | Score |
|-------|---------------------------------|-------|
| 1 | 5RM -Bench press | |
| 2 | 5RM -Back squat | |
| 3 | Counter movement Jump | |
| 4 | Overhead medicine ball | |
| 5 | Shoulder Joint Flexibility Test | |
| 5 | Sit and reach Test | |
| 7 | Hand-Eye Coordination Test | |
| 8 | Tennis speed Test | |
| 9 | Tennis accuracy Test | |

## **Dynamic warm-up content**

(Athlete in Photo: One of the participants)

## 1. High-knee walk

While walking, lift knee towards chest, raise body on toes, and swing alternating arms.





### 2. Straight-leg march

Straight-leg march. While walking with both arms extended in front of body, lift one extended leg towards hands then return to starting position before repeating with other leg.





### 3. Hand walk

With hands and feet on the ground and limbs extended, walk feet towards hands while keeping legs extended then walk hands forward while keeping limbs extended.





## 4. Lunge walks.

Lunge walks. Lunge forward with alternating legs while keeping torso vertical.



## 5. Backward lunge.

Move backwards by reaching each leg as far back as possible.



## 6. High-knee skip.

While skipping, emphasize height, highknee lift, and arm action.





## 7. Lateral shufflfle.

Move laterally quickly without crossing feet.



## 8. Back pedal.

While keeping feet under hips, take small steps to move backwards rapidly.



## 9. Heel-ups.

Rapidly kick heels towards buttocks while moving forward.



# 10. High-knee run.

Emphasize knee lift and arm swing while moving forward quickly.



# **Training content**

(Athlete in Photo: One of the participants)

Unilateral resistance training content

**Unilateral Bench Press Dumbbell** 





VIPR energy barrel for unilateral bench press









Bulgarian Heel Lift



One-handed push-ups on box





medicine ball forward throw



Self-weighted cross lunge jump





Single foot hurdle vertical jump



# Unilateral resistance training content

### **Bench Press for Dumbbell**





#### VIPR energy barrel for bench press





### Bilateral Weight Squat





Bulgarian Heel Lift





High five with push-ups





Double-sided medicine ball forward throw





#### Jump box



**Hurdle Vertical Jump** 





# Statistical Analysis Plan

| | Interven<br>tion | Pre | Post-1 | Post-2 | Δ | Statistical Analysis | |
|---|---|---|---|---|---|---|---|
| Grouping of subjects | | | | | | T-test/ANOVA | ANOVA |
| | | | | | | Within group | between groups |
| Subject-1 | $X_{\mathrm{U}}$ | $X_UO_1$ | $X_UO_2$ | $X_{\mathrm{U}}\mathrm{O}_{3}$ | Post1-pre $(O_{\Delta 1})$<br>Post2-pre $(O_{\Delta 2})$<br>Post2-Post1 $(O_{\Delta 3})$ | Post1 VS pre (T-test) Post2 VS pre (T-test) Post2 VS Post1 (T-test) O $_{\Delta 1}$ VS O $_{\Delta 2}$ VS O $_{\Delta 3}$ (ANOVA) | Post-1: $O_{\Delta 1} \text{ VS } O_{\Delta 4} \text{ VS } O_{\Delta 7} \text{ VS } O_{\Delta 10}(\text{ANOVA})$ Post-2: $O_{\Delta 2} \text{ VS } O_{\Delta 5} \text{ VS } O_{\Delta 8} \text{ VS } O_{\Delta 11}(\text{ANOVA})$ |
| Subject-2 | $X_{\mathrm{B}}$ | $ m X_BO_4$ | $X_BO_5$ | $X_{ m B}{ m O}_6$ | Post1-pre $(O_{\Delta 4})$<br>Post2-pre $(O_{\Delta 5})$<br>Post2-Post1 $(O_{\Delta 6})$ | Post1 VS pre (T-test) Post2 VS pre (T-test) Post2 VS Post1 (T-test) O <sub>Δ4</sub> VS O <sub>Δ5</sub> VS O <sub>Δ6</sub> (ANOVA) | |
| Subject-3 | X <sub>C</sub> | X <sub>C</sub> O <sub>7</sub> | X <sub>C</sub> O <sub>8</sub> | $X_CO_9$ | Post1-pre $(O_{\Delta7})$<br>Post2-pre $(O_{\Delta8})$<br>Post2-Post1 $(O_{\Delta9})$ | Post1 VS pre (T-test) Post2 VS pre (T-test) Post2 VS Post1 (T-test) O <sub>Δ7</sub> VS O <sub>Δ8</sub> VS O <sub>Δ9</sub> (ANOVA) | |
| CG | X | XO <sub>10</sub> | XO <sub>11</sub> | XO <sub>12</sub> | $\begin{array}{ccc} Post1\text{-pre} & (O_{\Delta 10}) \\ Post2\text{-pre} & (O_{\Delta 11}) \\ Post2\text{-Post1}(O_{\Delta 12}) \end{array}$ | Post1 VS pre (T-test) Post2 VS pre (T-test) Post2 VS Post1 (T-test) O $_{\Delta 10}$ VS O $_{\Delta 11}$ VS O $_{\Delta 12}$ (ANOVA) | |

#### Reference

- Speirs, D. E., Bennett, M. A., Finn, C. V., & Turner, A. P. (2016). Unilateral vs. bilateral squat training for strength, sprints, and agility in academy rugby players. The Journal of Strength & Conditioning Research, 30(2), 386-392.
- Davó, J. L. H., Jiménez, P. M., & Solana, R. S. (2018). Comparison of six weeks eccentric overload training between bilateral and unilateral squat in basketball players. European Journal of Human Movement, 40, 111-121.
- Ramírez-Campillo, R., Burgos, C. H., Henríquez-Olguín, C., Andrade, D. C., Martínez, C., Álvarez, C., ... & Izquierdo, M. (2015). Effect of unilateral, bilateral, and combined plyometric training on explosive and endurance performance of young soccer players. The Journal of Strength & Conditioning Research, 29(5), 1317-1328.
- Ji, S., Donath, L., & Wahl, P. (2022). Effects of alternating unilateral vs. bilateral resistance training on sprint and endurance cycling performance in trained endurance athletes: A 3-armed, randomized, controlled, pilot trial. The Journal of Strength & Conditioning Research, 36(12), 3280-3289.
- Faigenbaum, A. D., Bellucci, M., Bernieri, A., Bakker, B., & Hoorens, K. (2005).

  ACUTE EFFECTS OF DIFFERENT WARM-UP PROTOCOLS ON

  FITNESS PERFORMANCE IN CHILDREN
- Faigenbaum, A. (2009). Youth resistance training. Colorado Springs: NSCA Hot Topic

Series.

- Carter, J., & Greenwood, M. (2014). Complex training reexamined: Review and recommendations to improve strength and power. Strength & Conditioning Journal, 36(2), 11-19.
- Fernandez-Fernandez, J., Ellenbecker, T., & Ulbricht, A. (2013). Effects of a 6-week junior tennis conditioning program on service velocity. Journal of sports science & medicine, 12(2), 232.
- Ignjatovic, A. M., Markovic, Z. M., & Radovanovic, D. S. (2012). Effects of 12-week medicine ball training on muscle strength and power in young female handball players. The Journal of Strength & Conditioning Research, 26(8), 2166-2173.